CLINICAL TRIAL: NCT04521556
Title: Is Postoperative Quality of Recovery After Unilateral Nephrectomy Related to the Type of Anesthesia and Analgesia?
Brief Title: Effect of Epidural Anesthesia and Analgesia on Quality of Recovery After Unilateral Nephrectomy.
Acronym: QoR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of Split (Other)
Responsible Party: Principal Investigator, Ruben Kovac, Principal Investigator, University Hospital of Split
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2181-147-01/06/M.S.-19-2.
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia; Anesthesia Recovery Period; Nephrectomy; Patient Satisfaction; Postoperative Period; Quality of Life; Analgesia; Epidural
Keywords: general anesthesia; combined light general and epidural anesthesia; health related quality of life; nephrectomy
MeSH Terms: conditions — Patient Satisfaction; Agnosia | interventions — Anesthesia, Epidural; Analgesia, Epidural; Morphine; Ropivacaine; Anesthesia, General

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural anesthesia and analgesia (Active Comparator): Epidural catheter insertion: Th 9 - Th 10 or Th 10 - Th 11 using the midline approach.
  Safety of the epidural catheter was confirmed with lidocaine 60 mg. Epidural loading dose was given according to our classification (3,4,5 or 6 ml).
  Postoperative period in urology high care unit. Epidural analgesia ropivacaine/morphine was administered by a urologist according to our classification (2x2 ml, 2x3 ml and 3x3 ml).
  Interventions: Procedure: Epidural anesthesia with light general anesthesia; Procedure: Postoperative epidural analgesia
- Balanced general anesthesia and tramadol analgesia (Active Comparator): Postoperative period in urology high care unit.
  Interventions: Procedure: General anesthesia; Drug: Continuous intravenous analgesia

INTERVENTIONS:
Procedure: Epidural anesthesia with light general anesthesia — Epidural anaesthesia: mixture of ropivacaine 6.5 mg/ml and fentanyl 8.3 μg/ml.
  Light general anesthesia: isoflurane in mixture of 50/50 of nitrous oxide and oxygen to achieve Minimum alveolar concentration between 0.6 and 0.8.
  Arms: Epidural anesthesia and analgesia
Procedure: Postoperative epidural analgesia — Before the end of operation was given 4 ml of the mixture of ropivacaine 4.4 mg/ml and morphine 0.8mg/ml. Epidural analgesia was continued for next 24 hours with a mixture of ropivacaine 2.2 mg/ml and morphine 0.4 mg/ml.
  Other Names: Epidural analgesia with morphine and ropivacaine
  Arms: Epidural anesthesia and analgesia
Procedure: General anesthesia — Maintaining general anesthesia: nitrous oxide and oxygen in mixture 50/50 and isoflurane to achieve minimum alveolar concentration between 0.8 and 1.
  Fentanyl loading dose: 6-8 μg/kg. Additional fentanyl doses were given incrementally.
  Arms: Balanced general anesthesia and tramadol analgesia
Drug: Continuous intravenous analgesia — Tramadol 100 mg in the first hour followed by tramadol 300 mg continuously for the next 24 hours.
  Other Names: Continuous tramadol analgesia
  Arms: Balanced general anesthesia and tramadol analgesia

SUMMARY:
Different modality of anesthesia and analgesia could influence a postoperative quality of recovery (QoR). This study is exploring early QoR after unilateral nephrectomy in the two groups of anesthesia. The first group had a light general anesthesia with thoracic epidural anesthesia and postoperative epidural analgesia with morphine and ropivacaine. The second group had general anesthesia and a continuous postoperative analgesia with tramadol. The postoperative QoR was evaluated 24 hours after surgery.

DETAILED DESCRIPTION:
All participants were premedicated with diazepam 5 mg 12 hours and 1 hour before surgery. Thromboprophylaxis ( 4,000 - 6000 IU) depending on the body weight was given at least 12 hours before surgery. All participants were warmed to prevent unintended hypothermia. Participants were allocated by permuted-block randomisation into one of two groups: general anesthesia group and epidural anesthesia. The randomisation list was obtained from R program version 3.5.3. The group allocations were contained in a closed envelope that were opened before surgery after the completed enrollment procedure. All patients and infusions were wormed to prevent unintended hypothermia. Induction of general anesthesia was with midazolam 2.5 mg, fentanyl 100 μg, propofol 1-2 mg/kg and vecuronium 0.1 mg/kg.

Balanced crystalloid fluids were used to treat hypovolemia. Additionally, 6% Hydroxyethyl starch was used before blood transfusion products to treat profound hypovolemia.

Blood transfusions were given according to clinical situation. Bradycardia was treated with atropine. Hypotension was treated with ephedrine boluses. Anti-inflammatory drug metamizole (dipyrone) 2.5 g was given intravenously before the end of the surgery and after 12 hours after the surgery. Neostigmine 2.5 mg with atropine 1 mg was used for the reversal of the effects of non-depolarizing neuromuscular blocking agents after surgery. Participants were placed for one day in a urology high care unit provided with constant and vigilant nurse care.

Crystalloid infusions were used for maintaining diuresis. Gastroprotection was done with pantoprazole 40 mg. Metoclopramid 10 mg was given for postoperative nausea and vomiting (PONV).

The postoperative QoR was evaluated with three QoR scales. Scales for pain, anxiety and PONV were also examined. The 36-Item Short Form Survey (SF-36) questionnaire evaluated quality of life one month before and one month after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective radical nephrectomy
* American Society of Anesthesiologists (ASA) physical status classification system: I, II, III

Exclusion Criteria:

* Dementia
* Delirium
* Acute psychosis
* Emergent surgery
* Hospitalisation in Intensive care unit
* American Society of Anesthesiologists (ASA) physical status classification system: IV
* Reoperations
* Muscular diseases
* Montreal cognitive test <24 points
* Contraindications for epidural anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale of quality of recovery (QoR) | 24 hours after surgery
  Patient rated visual analog scale is a simple scale for rating the quality of recovery by placing "X" on the line. Poor recovery is on the left side of the line. Under the end of the left line is an explanation of poor recovery: in severe pain, nausea & vomiting, confused, immobilized, unable to eat and unable to communicate. Excellent recovery is on the right side of the line. Under the end of the line is a written explanation: without any pain, comfortable, alert, active, enjoying food and communicating freely.
Quality of recovery 40 (QoR-40) | 24 hours after surgery
  The QoR-40 measures five related dimensions of quality of recovery: emotional state (8 items), physical comfort (12 items), physical independence (5 items), psychological support (7 items) and pain (7 items). Each item is rated on a 5 point Likert scale. Minimal possible score is 40 and maximal possible score is 200.
Quality of recovery 15 (QoR-15) | 24 hours after surgery
  Quality of recovery (QoR-15) is a short version of QoR - 40 questionnaire. The QoR-15 questionnaire has 15 items scaled from 0 to 10. Minimum score is 0, and maximum 150. It is shorter, user friendly and less time consuming then extensive QoR-40 questionnaire.

SECONDARY OUTCOMES:
Visual analog scale of pain- at rest and during coughing and straining | 24 hours after surgery
  Patient rated visual analog pain scale is a simple scale for rating the quality of recovery by placing "X" on the line. No pain at all is written on the left side of the line. The worst possible pain is on the right side of the line.
Numerical pain scale - at rest and during coughing and straining | 24 hours after surgery
  Similar to the visual analog scale of pain, but instead of line, it consists of a sequence of numbers (0-10). For some participants, scaling pain in numbers (0-10) is more clear than analog scale.
Visual pain scale with faces- at rest and during coughing and straining | 24 hours after surgery
  Similar to the numeric pain scale. If pain scaling in numbers is vaguely, then six faces with emotional expression ranging from a happy smiling to a crying face with tears explain numbers under the faces (0,2,4,6,8,10).
Visual analog scale of anxiety | 24 hours after surgery
  Patient rated visual analog scale is a simple scale for rating the level of anxiety by placing "X" on the line. No anxiety at all is written on the left side of the line. The worst possible anxiety is on the right side of the line.
Numerical anxiety scale | 24 hours after surgery
  Similar to the visual analog scale of anxiety, but instead of line, it consists of a sequence of numbers (0-10). For some participants, scaling in numbers (0-10) is more clear than analog scale.
Visual anxiety scale with faces | 24 hours after surgery
  Similar to the numerical anxiety scale. For some patients quantifying pain in numbers is vague, but if they can observe faces with different emotional expressions ranging from a happy smiling to a crying face with tears. Under the faces are written corresponding numbers (0,2,4,6,8,10)
The short form health survey version one (SF-36:I) | 24 hours after surgery and one month after surgery
  The short form health survey version one (SF-36:I.) measure eight dimensions of quality of life: physical functioning (10 items), role limitation due to physical problems (4 items), bodily pain (2 items), social functioning (2 items), mental health (5 items), role limitation due to emotional problems (3 items), vitality (4 items) and general health perception (5 items). Each dimension has a possible score of 0 (poor health) to 100 (excellent health).
Simplified postoperative nausea and vomiting (PONV) impact scale | 24 hours after surgery
  PONV impact scale consists of 2 questions that are scored from 0 to 3. Five points or six defines clinically important PONV.
Global visual analog and numeric scale of nausea intensity | 24 hours after surgery
  Scale for rating the nausea intensity by placing "X" on the line. No nausea at all is written on the left side of the line. The worst possible nausea experienced is on the right side of the line. Under the line are written numbers (0-10).

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Kovac, Principal Investigator — University Hospital Split, Department of Anesthesiology and Intensive Care; Bozidar Duplancic, Study Director — University Hospital Split, Department of Anesthesiology and Intensive Care; Verica Ilijev, Study Chair — University Hospital Split, Department of Anesthesiology and Intensive Care; Ivo Juginovic, Study Chair — University Hospital Split, Department of Urology; Ivan Velat, Study Chair — University Hospital Split,Department of Urology; Hrvoje Vucemilovic, Study Chair — University Hospital Split, Department of Anesthesiology and Intensive Care; Svjetlana Dosenovic, Study Chair — University Hospital Split, Department of Anesthesiology and Intensive Care
Locations (1):
- University Hospital Split, Split, Croatia

REFERENCES:
- [Background] Greg Snow (2020) blockrand: Randomization for Block Random Clinical Trials. R package version 1.5. https://CRAN.R-project.org/package=blockrand
- [Background] Stamer UM, Hothker F, Lehnen K, Stuber F. [Postoperative analgesia with tramadol and metamizol. Continual infusion versus patient controlled analgesia]. Anaesthesist. 2003 Jan;52(1):33-41. doi: 10.1007/s00101-002-0427-1. German. PMID 12577163
- [Background] Myles PS. Measuring quality of recovery in perioperative clinical trials. Curr Opin Anaesthesiol. 2018 Aug;31(4):396-401. doi: 10.1097/ACO.0000000000000612. PMID 29846193
- [Background] Gornall BF, Myles PS, Smith CL, Burke JA, Leslie K, Pereira MJ, Bost JE, Kluivers KB, Nilsson UG, Tanaka Y, Forbes A. Measurement of quality of recovery using the QoR-40: a quantitative systematic review. Br J Anaesth. 2013 Aug;111(2):161-9. doi: 10.1093/bja/aet014. Epub 2013 Mar 6. PMID 23471753
- [Background] Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br J Anaesth. 2000 Jan;84(1):11-5. doi: 10.1093/oxfordjournals.bja.a013366. PMID 10740540
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134
- [Background] Kleif J, Gogenur I. Severity classification of the quality of recovery-15 score-An observational study. J Surg Res. 2018 May;225:101-107. doi: 10.1016/j.jss.2017.12.040. Epub 2018 Feb 21. PMID 29605019
- [Background] Cao X, Yumul R, Elvir Lazo OL, Friedman J, Durra O, Zhang X, White PF. A novel visual facial anxiety scale for assessing preoperative anxiety. PLoS One. 2017 Feb 14;12(2):e0171233. doi: 10.1371/journal.pone.0171233. eCollection 2017. PMID 28196099